CLINICAL TRIAL: NCT00552773
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Group Trial of Cyclamen Europaeum Extract Nasal Spray 10% (v/v) in the Treatment of Subjects With Acute Sinusitis
Brief Title: Pilot Study to Determine Efficacy of Cyclamen Europaeum Extract Nasal Spray in Patients With Acute Sinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 434-083
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2011-11

CONDITIONS: ACUTE SINUSITIS
Keywords: SINUSITIS; CYCLAMEN
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclamen Europaeum (Experimental)
  Interventions: Drug: Cyclamen Europaeum
- Placebo (Placebo Comparator)
  Interventions: Drug: Cyclamen Europaeum

INTERVENTIONS:
Drug: Cyclamen Europaeum — Nasal spray 10% (V/V),one spray per nostril daily for 7 days.

SUMMARY:
To evaluate the efficacy and safety of Cyclamen europaeum extract 10 % (v/v) compared to placebo in subjects with acute sinusitis

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18-70
2. Must be symptomatic on the basis of subject assessments of total sympton score.
3. Evidence of mucopurulence on nasal endoscopy
4. Evidence of inflammation upon nasal endoscopy
5. CT scan with radiographic signs of acute sinusitis
6. Able to complete all study activities or procedures through the end of the study, including all visits and tests, and capable of selfadministration of study medication
7. Agree to abide by the study protocol and its restrictions

Exclusion Criteria:

1. Known history of hypogammaglobulinemia, immotile cilia syndrome, atrophic rhinitis, rhinitis medicamentosa, or cystic fibrosis
2. Known hypersensitivity to Cyclamen, Primula, or other Primulaceae
3. Serious unstable comorbidity such as malignancy (other than squamous or basal cell carcinoma of the skin) or sever renal or hepatic disease.
4. Abnormal screening laboratory/imaging test results
5. Condition(s) that compromise the ability to either administer the agent or assess the risks/benefits (eg mucocele, choanal polyp, Stage 4 polyposis or cyst extending below the inferior turbinate, deviated septum, facial trauma, or birth defect)
6. Expansile mass or bony erosion on sinus radiograph
7. Females who are pregnant, planning to become pregnant or currently breastfeeding.
8. History of viral upper respiratory infection (URI) in the past 2 weeks
9. Temperature greater than 102.5°F
10. Facial or periorbital edema
11. Local complications including orbital cellulitis; acute abnormalities of extraocular movements; cavernous vein thrombosis; dental or facial abscess
12. Altered mental status
13. Recent nasal or sinus surgery (within 3 months or less) or planned surgery within the next 3 months
14. Use of intranasal antibiotics within the previous 30 days or systemic antibiotics within the previous 15 days
15. Use of oral and/or topical nasal decongestants within the previous 7 days
16. Had radiation therapy or chemotherapy within the previous 12 months
17. Have used an investigational drug or device within 30 days prior to screening
18. Have a history of illegal drug or alcohol abuse within the past 5 years
19. Have major unstable organ system disease that could place the subject at increased risk of complications, interfere with study participation, or confound any of the study objectives Subjects who have asthma, seasonal and/or perennial allergic rhinitis will be allowed to enter the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Subjective: The mean change in Total Symptom Score (TSS). Objective: The mean change in the percent of sinus occlusion as determined by CT scans. | 1 year

SECONDARY OUTCOMES:
TSS change from Baseline to each post-dose visit for each symptom scoring Change from Baseline for the individual symptom scores Time to cure rate Frequency of acute sinusitis episodes The presence/absence of mucopurulence and inflamed nasal mucosa | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Barreto, MD, Principal Investigator — Memorial Clinical Reasearch, OK
Locations (25):
- United States (25):
  - Alliance Clinical Research, Birmingham, Alabama
  - Center of Research Excellence, LLC, Oxford, Alabama
  - Clinical Research Connections, Jonesboro, Arkansas
  - Southeast Clinical Research, Gainsville, Florida
  - Orlando Rangel, MD, PA, Tampa, Florida
  - Premier Health Research Center, Winter Haven, Florida
  - Peak Medical Research, LLC, Owensboro, Kentucky
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Las Vegas Physicians Research Group, Henderson, Nevada
  - LAND Clinical Studies, LLC, West Caldwell, New Jersey
  - Health Science Research Center, Cortland, New York
  - Medical Research Associates of Central ew York, PLLC, North Syracuse, New York
  - American Institute of Healthcare and Fitness Clinical Research, Raleigh, North Carolina
  - Jones Family Pratice, Shelby, North Carolina
  - Memorial Clinical Research, Oklahoma City, Oklahoma
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - ADAC Research, PA, Greenville, South Carolina
  - Carolina Research, Orangeberg, South Carolina
  - Austin Ear, Nose and Throat Clinic, Austin, Texas
  - West Lake Ffamily Practice/Time Point Clinical Research, Austin, Texas
  - San Antonio Ear, Nose & Throat Research, San Antonio, Texas
  - Live Oak Allergy and Asthma Clinic, San Antonio, Texas
  - Clinical Health Research LLC, Sugar Land, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Virginia Adult and Pediatric Allergy and Asthma, PC, Richmond, Virginia